CLINICAL TRIAL: NCT02368561
Title: A Pilot Study of the Effects of 3 Retro-calcaneal Hyalin G-F 20 Injection on the Clinical and Radiological Changes in 20 Adult Patients With Changes in Insertional Achilles Tendinopathy.
Brief Title: Treatment of Insertional Achilles Tendinopathy by Hyaluronic Acid Injection
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC140082CTIL
Record Dates: First submitted 2015-02-02; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2014-12

CONDITIONS: Insertional Achilles Tendinitis
MeSH Terms: interventions — hylan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyaluronic Acid Injection (Experimental): Hyaluronic Acid Injection in 20 adult patients with IAT
  Interventions: Drug: Injection of Hyaluronic Acid -" SYNVISC" (hylan G-F 20)

INTERVENTIONS:
Drug: Injection of Hyaluronic Acid -" SYNVISC" (hylan G-F 20) — US guided weekly injection of sodium hyaluronate administered for 3 week in adult subjects with insertional achilles tendinopathy

SUMMARY:
A pilot study of the effects of 3 retro-calcaneal hyalin G-F 20 injection on the clinical and radiological changes in 20 adult patients with changes in insertional achilles tendinopathy.

DETAILED DESCRIPTION:
Pain of the achilles tendon commonly affects young active patients, with lifetime incidence that may be as high as 40 to 50 percent in competitive athletes. About 20% of the achilles tendinopathy injuries occur in the insertion point of the achilles tendon into the calcaneus bone1. The leading theories for the mechanism of the disorder are inflammatory response or mechanical tendon overuse. Still, the exact pathogenesis of Insertional Achilles tendinitis (IAT) is unclear, and as so the conservative management of IAT is less successful than the management of the Non-insertional tendinopathy. Previous histological description, in an unpublished data of the insertion point showed that the main pathologic features were found to be in the bone and cartilage tissues. The achilles tendon, in those studies, was almost intact. The histological features of the cartilage tissue were advanced degenerative changes, which resemble the pathologic changes of Osteoarthritis. This observation encourages to try treating IAT with management strategies that showed to be beneficial in OA( OsteoArthritis). One of the more acceptable non-surgical methods in treating osteoarthritis is intra-articular viscosupplementation injection. The investigators hypothesis, based on the histopathological finding, is that viscosupplementation may be a therapeutic option also for individuals with IAT. The purpose of this study is to show the impact of Hyalin G-F 20 injection in patients with Insertional Achilles tendinitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with chronic (>6 months) posterior heel pain localized above the insertion point of the achilles tendon with evidence of IAT in ankle X-RAY and MRI.

Exclusion Criteria:

1. Previous surgical treatment.
2. Previous HA(Hyaluronic Acid), PRP (Platelet Rich Plasma) or steroids injection in the last 6 months.
3. Previous two or more steroids injection.
4. Plantaris muscle injury.
5. Posterior ankle impingement.
6. Achilles tendon rapture.
7. Previous calcaneal fracture

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-01 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change in the VISA-A questionnaire score | Change in the VISA-A questionnaire score during 6 months follow-up
  The VISA-A questionnaire score at 3 points during the follow-up: before the treatment, one month after the procedure and 6 months from the procedure.

SECONDARY OUTCOMES:
The sonographic signs | Change in the achilles tendinosis sonographic signs during 6 months follow-up
  The sonographic signs in the achilles enthesis- hypoechoic swelling, hyperemia, peritendinitis, fluid in the retrocalcaneal bursa, osseous prominence at the posterosuperior calcaneus.

CONTACTS AND LOCATIONS:
Overall Officials: Meir Nyska, Prop, Study Director — head of orthopedic department

REFERENCES:
- [Background] Roche AJ, Calder JD. Achilles tendinopathy: A review of the current concepts of treatment. Bone Joint J. 2013 Oct;95-B(10):1299-307. doi: 10.1302/0301-620X.95B10.31881. PMID 24078523
- [Background] Wiegerinck JI, Kerkhoffs GM, van Sterkenburg MN, Sierevelt IN, van Dijk CN. Treatment for insertional Achilles tendinopathy: a systematic review. Knee Surg Sports Traumatol Arthrosc. 2013 Jun;21(6):1345-55. doi: 10.1007/s00167-012-2219-8. Epub 2012 Oct 6. PMID 23052113
- [Background] Oshri Y, Palmanovich E, Brin YS, Karpf R, Massarwe S, Kish B, Nyska M. Chronic insertional Achilles tendinopathy: surgical outcomes. Muscles Ligaments Tendons J. 2012 Sep 10;2(2):91-5. Print 2012 Apr. PMID 23738280
- [Background] Irwin TA. Current concepts review: insertional achilles tendinopathy. Foot Ankle Int. 2010 Oct;31(10):933-9. doi: 10.3113/FAI.2010.0933. No abstract available. PMID 20964977
- [Background] Kearney R, Costa ML. Insertional achilles tendinopathy management: a systematic review. Foot Ankle Int. 2010 Aug;31(8):689-94. doi: 10.3113/FAI.2010.0689. PMID 20727317
- [Background] Petrou MJ. Re: Kuipers H, Ruijsch van Dugteren G. Letter to the editors - the prohibited list and cheating in sport. Int J Sports Med 2006; 27: 80 - 82. Int J Sports Med. 2006 Jan;27(1):83-4. doi: 10.1055/s-2005-873070. No abstract available. PMID 16388448
- [Background] Kumai T, Muneta T, Tsuchiya A, Shiraishi M, Ishizaki Y, Sugimoto K, Samoto N, Isomoto S, Tanaka Y, Takakura Y. The short-term effect after a single injection of high-molecular-weight hyaluronic acid in patients with enthesopathies (lateral epicondylitis, patellar tendinopathy, insertional Achilles tendinopathy, and plantar fasciitis): a preliminary study. J Orthop Sci. 2014 Jul;19(4):603-11. doi: 10.1007/s00776-014-0579-2. Epub 2014 May 10. PMID 24817495